CLINICAL TRIAL: NCT00386906
Title: Sentinel Lymph Node Localization and Biopsy for Conjunctival and Eyelid Melanoma
Brief Title: Sentinel Lymph Node (SLN) Biopsy for Conjunctival/Eyelid Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GSP00-106; NCI-2012-01480 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Eye Disease; Melanoma
Keywords: Melanoma; Conjunctival Melanoma; Malignant Melanoma of the Conjunctiva; Malignant Melanoma of the Eyelid; Sebaceous Cell Carcinoma; Sebaceous Cell Carcinoma of the Conjunctiva; Sebaceous Cell Carcinoma of the Eyelid; Sentinel Lymph Node; Lymphatic Mapping; Eyelid; Eyelid Lesion
MeSH Terms: conditions — Eye Diseases; Melanoma | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentinel Lymph Node (SLN) Biopsy (Other): Intraoperative lymphatic mapping, then biopsy/removal of the conjunctiva/eyelid tumor.
  Interventions: Procedure: Sentinel Lymph Node Mapping and Biopsy

INTERVENTIONS:
Procedure: Sentinel Lymph Node Mapping and Biopsy — Intraoperative lymphatic mapping, then biopsy/removal of the conjunctiva/eyelid tumor.

SUMMARY:
The goal of this clinical research study is to find the sentinel lymph node (SLN) (s) and biopsy it (them) to see if the patient has small or low volume metastatic disease that would otherwise have been missed.

DETAILED DESCRIPTION:
You have had your conjunctival or eyelid tumor surgically removed or it is scheduled to have it removed. You will have lymphatic mapping before the tumor is removed. Lymphatic mapping is when a small volume of Tc99m-Sulfur colloid is injected by an ophthalmologist after which some radiologic images are taken.

If you are able to become pregnant, blood (about 2 teaspoons) will be drawn for a pregnancy test, within 7 days before the biopsy. To take part in this study, you must not be pregnant.

You will then go to the operating room and have intraoperative SLN mapping and biopsy. If the SLN is positive on permanent section, you will go on to have complete lymph node dissection, which involves removal of all the lymph nodes around the positive SLN. Then the disease will be restaged and you may require further treatment after consultation with their oncologist.

Your medical record will be reviewed, and information from your medical record will be recorded and reviewed to help researchers better identify those patients who have microscopic lymph node disease. The information collected from your medical records will include information about your sex, age, what type of cancer that you have, as well as the size of the cancer and its location.

Researchers hope to identify those patients who have microscopic lymph node disease before it becomes clinically obvious. With this technique, researchers could potentially identify occult metastatic disease which would otherwise go unnoticed until it was too advanced. Patients in this study will have to see the ophthalmologist every three months and have the usual metastatic workup, which is routine for conjunctival/eyelid melanoma.

Length of Study:

Your active participation on this study will be over once the biopsy is over. You will continue to be observed on study for 5 years after the biopsy.

Long-Term Follow-Up:

Every 3 months for the first year after the biopsy, and every 6 months after that until 5 years after the biopsy, you will have an eye exam to check the status of the disease.

Every 6 months for the first year after the biopsy, blood (less than 1 teaspoon) will be drawn for liver function tests. You will also have a chest x-ray. You will then have these tests 1 time each year for 5 years after the biopsy.

You will have a head and neck CT or MRI every 6 months for the first year after the biopsy to make sure the disease has not come back. The head and neck CT or MRI will be repeated 1 time each year for 5 years after the biopsy.

This is an investigational study. A total of 38 patients will take part in this study. All will be enrolled at MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 years of age or older.
2. Histologically documented malignant melanoma of the conjunctiva/eyelid greater than or equal to 1 millimeter in thickness, or those less than 1 mm thick that have evidence of ulceration, mitotic figures or are Clark IV.
3. A CXR, liver enzymes, and a head and neck computed tomography (CT) or magnetic resonance imaging (MRI) negative for evidence of metastasis.
4. Participant must have a negative ultrasound of regional lymph nodes (i.e., within 6 weeks of study enrollment).
5. Patient provided written informed consent. In the event that non-English speaking participants are eligible for this study, a short form (if applicable) or an ICD in their language, will be utilized and completed in accordance with the MDACC Policy for Consenting Non-English Speaking Participants.

Exclusion Criteria:

1) Pregnant or nursing females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2000-05-30 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Sentinel Lymph Node (SLN) Positivity in Conjunctival/eyelid Melanomas | 3 months
  The frequency of lymphatic drainage basins for bulbar versus palpebral conjunctiva and for nasal and the temporal quadrants estimated with 95% confidence intervals. The rate of identification of SLN evaluated with a confidence interval. The probability of positive SLN in primary conjunctival and eyelid melanoma estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Bita Esmaeli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org